CLINICAL TRIAL: NCT07328685
Title: Examining the Effectiveness of Basic Body Awareness Therapy in Individuals With Migraine
Brief Title: Basic Body Awareness Therapy in Individuals With Migraine
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Yasemin KARAASLAN, Principal Investigator, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HMKU-BBAT-2026
Record Dates: First submitted 2025-12-27; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Migraine
Keywords: migraine; functional status; sleep; quality of life
MeSH Terms: conditions — Migraine Disorders | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Body Awareness Therapy Plus Standard Treatment (Experimental): Participants in this group will receive body awareness therapy in addition to standard treatment. The exercise program will be implemented twice over an eight-week period.
  Interventions: Behavioral: Exercise; Behavioral: Standart therapy
- Standart Treatment (Active Comparator): Participants in this group will receive standard treatment without the additional body awareness therapy.
  Interventions: Behavioral: Standart therapy

INTERVENTIONS:
Behavioral: Exercise — Participants will receive body awareness therapy. The program will be administered over an eight-week period and will include exercises appropriate for the study population.
  Arms: Body Awareness Therapy Plus Standard Treatment
Behavioral: Standart therapy — Standard treatment will be in the form of individual information sessions lasting approximately 30 minutes for both groups. Brochures will be created for distribution to individuals.

SUMMARY:
One biopsychosocial approach proven effective in headache treatment is basic body awareness therapy. This study was planned to evaluate the effectiveness of basic body awareness training and lifestyle recommendations in individuals diagnosed with migraine. Functional status will be assessed using the Migraine-Related Disability Assessment Scale (MIDAS), sleep quality using the Jenkins Sleep Scale (JUS), and quality of life using the Headache Impact Test. Assessment of functional status, sleep quality, and quality of life will be performed before treatment and after treatment (at the end of week 8).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with migraine,
* Experiencing at least 3 migraine attacks per month,
* Between the ages of 18 and 55 and who volunteer to participate in the study.

Exclusion Criteria:

* History of secondary headaches,
* Being pregnant,
* Having any other neurological disease besides migraine,
* Having other secondary headaches in addition to migraine,
* History of malignancy,
* Regularly practicing meditation, yoga, or mindfulness-based practices.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Pain Diary | Individuals will be asked to regularly complete a pain diary during the 4-week period before the program, during the program, and during the 4-week follow-up period after the training is completed.
  The severity, duration, and frequency of headaches during attacks will be recorded daily by the participants.

SECONDARY OUTCOMES:
Functional status | Baseline and at the end of the 8-week intervention
  The Migraine Disability Assessment Scale will be used to determine the functional status associated with migraine.
Sleep quality | Baseline and at the end of the 8-week intervention
  Individuals' sleep quality will be assessed using the Jenkins Sleep Scale.
Quality of life related to headaches. | Baseline and at the end of the 8-week intervention
  The Headache Impact Test will be used to assess the impact of headache on quality of life.

IPD SHARING:
Plan to Share IPD: No